



Participant identification number:

## Mr Daniel Howgate

Study Code:

Honorary Specialty Registrar Trauma & Orthopaedic Surgery and DPhil Student Botnar Institute of Musculoskeletal Sciences, University of Oxford, Old Road, Oxford, OX3 7LD

E-mail: daniel.howgate@ndorms.ox.ac.uk Oxford telephone number: 01865 760063

Site ID Code:

| SURGEON PARTICIPANT CONSENT FORM: CONSULTANTS & FELLOWS | | | | | |
|---|---|---|---|---|---|
| A prospective randomised controlled study assessing surgical performance and the impact of simulation training in primary THR | | | | | |
| Name of Researcher: | | | lf | you agree, please initial | box |
| 1. | I confirm that I have read the information sheet dated (version) for this study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason. | | | | |
| 3. | I understand that relevant sections of my anonymised data collected during the study may be looked at by individuals from University of Oxford, from regulatory authorities and from the NHS Trust(s), where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | | |
| 4. | 4. I agree to take part in this study. | | | | |
| Name of Participant | | <br>Date | | Signature | |
| Name of Person taking<br>Consent | | Date | | Signature | |

Surgeon Participant Consent form: Cons/AF THR Performance & Assessment Professor Jonathan Rees Version 2.0 12<sup>th</sup> October 2019 IRAS Project number: 270167 REC Reference number: 19/SC/0492

<sup>\*1</sup> copy for participant; 1 copy for researcher site file; 1 (original) to be kept in medical notes (if participant is a patient).